CLINICAL TRIAL: NCT02300662
Title: Early Mobilization With a Cycle Ergometer for Critical Patients on Invasive Mechanical Ventilation in the Intensive Care Unit (MoVe-ICU Study): Study Protocol for a Randomized Controlled Trial
Brief Title: Early Mobilization for Critical Patients on Invasive Mechanical Ventilation in the Intensive Care Unit
Acronym: MoVe-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-0530
Record Dates: First submitted 2014-10-30; First posted 2014-11-25 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cycle Ergometer (Experimental): Conventional physiotherapy and cycle ergometer 20 minutes, at 20 cycles per minute, once per day for as long as they remain on invasive mechanical ventilation
  Interventions: Device: Cycle Ergometer; Other: Conventional physiotherapy
- Conventional Physiotherapy (Sham Comparator): Upper and lower extremity functional diagonals from the proprioceptive neuromuscular facilitation method and manual bronchial hygiene exercises.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Device: Cycle Ergometer — Passive movement of the cycle ergometer will execute alternate flexions and extensions of the patients' knee and hips bilaterally for 20 minutes consecutively.
  Arms: Cycle Ergometer
Other: Conventional physiotherapy — Manual bronchial hygiene exercises: vibrocompression, manoeuvres with a manual resuscitator (bag squeezing) and aspiration of secretions where necessary.

SUMMARY:
A single blind randomized controlled trial (the MoVe ICU study) will be conducted to evaluate the effects on critical patients on invasive mechanical ventilation of early mobilization with a cycle ergometer.

DETAILED DESCRIPTION:
A single blind randomized controlled trial (the MoVe ICU study) will be conducted to evaluate the effects on critical patients on invasive mechanical ventilation of early mobilization with a cycle ergometer. Patients (age > 18 years) will be recruited for this study from among those admitted to the intensive care department at the Hospital de Clínicas de Porto Alegre. Eligible patients will have been on invasive mechanical ventilation for at least 24 to 48 hours, will have spent maximum of 1 week in hospital and will not exhibit any characteristics restricting lower extremity mobility. These subjects will be randomized to receive either conventional physiotherapy or conventional physiotherapy with an additional cycle ergometer intervention. The intervention will be administered passively for 20 minutes, at 20 revolutions per minute, once per day, throughout the time the patients remain on invasive mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* patients of both sexes aged >= 18 years will be recruited from among those admitted to the Hospital de Clínicas de Porto Alegre intensive care unit and put on invasive mechanical ventilation invasive mechanical ventilation for at least 24 to 48 hours after transfer from the emergency department or wards, no more than 1 week after admission

Exclusion Criteria:

* neuromuscular diseases causing motor deficits, such as strokes, multiple sclerosis, amyotrophic lateral sclerosis, myasthenia gravis and Guillain Barré syndrome.
* patients will also be excluded in the event of the following: extubation less than 48 hours after enrollment on the study
* haemodynamic instability (noradrenaline > 0.5 mc/kg/min for arterial blood pressure > 60 mmHg)
* complications during the protocol such as pneumothorax, deep vein thrombosis or pulmonary embolism
* Shilley catheter in the femoral vein
* reintubation
* delayed weaning (3 failed spontaneous ventilation tests)
* body mass index > 35 kg/m2
* emergence of eschar in the calcaneus area during the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
change in cross-sectional quadriceps thickness | baseline and after seven days of protocol
  ultrasound measurement of the vastus intermedius and the rectus femoris muscles thickness

SECONDARY OUTCOMES:
change in length of fascicle | baseline and after seven days of protocol
  ultrasound measurement of the length of fascicle
change in pennation angle of fascicles | baseline and after seven days of protocol
  ultrasound measurement of the pennation angle of fascicles
change in thickness of vastus lateralis muscle | baseline and after seven days of protocol
  ultrasound measurement of the thickness of vastus lateralis muscle
change in diaphragm thickness | baseline and after seven days of protocol
  ultrasound measurement of the diaphragm muscle thickness
change in diaphragm excursion | baseline and after seven days of protocol
  ultrasound measurement of the inspiratory and expiratory diaphragmatic excursion

CONTACTS AND LOCATIONS:
Overall Officials: Silvia R Vieira, ScD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] dos Santos LJ, de Aguiar Lemos F, Bianchi T, Sachetti A, Dall' Acqua AM, da Silva Naue W, Dias AS, Vieira SR. Early rehabilitation using a passive cycle ergometer on muscle morphology in mechanically ventilated critically ill patients in the Intensive Care Unit (MoVe-ICU study): study protocol for a randomized controlled trial. Trials. 2015 Aug 28;16:383. doi: 10.1186/s13063-015-0914-8. PMID 26314881